CLINICAL TRIAL: NCT06385990
Title: Clinical Study of the Efficacy and Safety of Utidelone (UTD1) Combined With Capecitabine as Adjuvant Therapy in Non-pCR Triple-negative Breast Cancer Patients After Neoadjuvant Therapy
Brief Title: Utidelone (UTD1) Plus Capecitabine in Non-pCR TNBC After Neoadjuvant Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024ks01
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: adjuvant chemotherapy; non-pCR
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UTD1 in combination with capecitabine (Experimental): UTD1 30mg / m², once a day on days 1-5; capecitabine: 1000mg / m², days 1-14, oral, twice / day; 21 days a treatment cycle of 6-8 cycles.
  Interventions: Drug: UTD1

INTERVENTIONS:
Drug: UTD1 — UTD1: 30mg / m², once a day on days 1-5; capecitabine: 1000mg / m², days 1-14, oral, twice / day; 21 days a treatment cycle of 6-8 cycles.
  Other Names: capecitabine

SUMMARY:
This trial is a multicenter, single-arm clinical trial to evaluate the efficacy and safety of UTD1 in combination with capecitabine for the adjuvant treatment of TNBC patients who did not achieve pathologic complete remission after neoadjuvant therapy. TNBC patients who did not achieve pathological complete remission or positive lymph node after neoadjuvant chemotherapy received adjuvant treatment with study drug.

Solution: UTD1 30mg / m², once a day on days 1-5; capecitabine: 1000mg / m², days 1-14, oral, twice / day; 21 days a treatment cycle of 6-8 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* 18 Years and older;
* Female;
* Breast cancer confirmed by pathological histology, ER-negative (<1% positive), PR-negative (<1% positive), and HER2-negative (IHC: HER2 (0), HER2 (1+), or HER2 (2+) and FISH non-amplification;
* Patients must receive full course of neoadjuvant chemotherapy before surgery and did not achieve pathological complete response (i. e., pathologically confirmed residual lesion, maximum diameter of 1cm) or / lymph node positive (ypN+);
* Previous neoadjuvant chemotherapy regimen included anthracycline, taxane, or a combination of both.
* Patients who clinically require radiotherapy of the affected breast or chest wall and regional lymph node area should receive radiotherapy before or after study medication;
* All toxicities related to previous antitumor therapy must return to Grade 1 (CTCAE v5.0), except alopecia;
* Within 1 week before enrollment, the blood routine examination was basically normal (taking the normal value of each study center as the standard): 1) Blood routine: hemoglobin (Hb) > 90g / L, White blood cell count (WBC) > 3.5*10^9 / L, Number of neutrophils (ANC) * 1.5*10^9 / L, Platelet count (PLT)* 100*10^9 / L; 2) Renal function: upper limit of normal serum creatinine value; 3) Liver function: for patients without liver metastasis: glutamulate aminotransferase (AST), glutamate aminotransferase (ALT), alkaline phosphatase (ALP) are less than 2.5 times of the upper limit of normal value, and totle bilirubin is less than 1.25 times of the upper limit of normal value; for patients with liver metastasis, AST, ALT, ALP, ALT, ALP, are less than 5 times of the upper limit of normal value, and totle bilirubin is less than 1.25 times of the upper limit of normal value;
* The ECOG physical status score for patients must be 0 or 1;

Exclusion Criteria:

* Metastatic breast cancer at diagnosis;
* Breast cancer patients who did not completed surgery;
* History of other malignancies within 5 years prior to randomization, but patients with the following tumors may participate in the study: carcinoma of the cervix in situ, colon in situ, melanoma in situ and basal cell carcinoma of the skin and squamous cell carcinoma;
* Any other non-malignant systemic disease (cardiovascular, renal, liver, etc.) that hinders the implementation or follow-up of the treatment program;
* Symptomatic congestive heart failure (New York Heart Association Grade II-IV), symptomatic or poorly controlled arrhythmia, history of congenital long QT syndrome or corrected QTc> 500ms at screening, history of uncontrolled hypertension or hypertensive crisis or hypertensive encephalopathy;
* History of interstitial pneumonia, Need for steroids or evidence of active pneumonia;
* Suffering from an active autoimmune disease, and required systemic treatment in the past 2 years (i. e., use of disease regulators, corticosteroids, or immunosuppressive drugs);
* Patients with a known infection with human immunodeficiency virus (HIV);
* Patients with active infections requiring systemic treatment;
* Any hormonal medication (such as raloxifene, tamoxifen, or other selective oestrogen receptor modulators) for osteoporosis or breast cancer prophylaxis (only patients who have discontinued these drugs before randomization may participate in the study);
* The patient received either capecitabine or utiderone before surgery;
* Pregnant or lactating women;
* Known or suspected allergy to any study drug or excipients;
* Prohibition of corticosteroids;
* Any other condition the investigator considers inappropriate to participate in the trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-03-29 (Estimated); Study Completion 2027-03-29 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival (DFS) | 2 years
  2-year DFS will be defined as the percentage of patients alive without recurrence or metastasis of disease at 2 years measured from the date of enrollment.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 2 years (from date of enrollment to the date of death).
  OS was calculated for each patient based on time of enrollment to time of death.
Disease Free Survival (DFS) | Up to 2 years (from date of surgery to the date of recurrence / metastasis).
  DFS was measured from surgery to the time of recurrence or metastasis.
Invasive Disease free survival (iDFS) | From the date of surgery to the time of invasive local, axillary or distant recurrence, invasive contralateral breast cancer or death from any cause (whichever occurs first)., up to 2 years.
  iDFS was measured from surgery to the time of invasive local, axillary or distant recurrence, invasive contralateral breast cancer or death from any cause (whichever occurs first).
Distant Disease-free Survival (DDFS) | From the date of surgery to distant recurrence, or death due to any cause (up to 2 years).
  DDFS is defined as the time from surgery to distant recurrence, or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Quchang Ouyang, Changsha, Hunan, China